CLINICAL TRIAL: NCT03747302
Title: HPV Message Testing and Social Media Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Norris Cotton Cancer Center (Other)
Responsible Party: Principal Investigator, Ardis Olson, MD, Physician, Professor of Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D18180; 3P30CA023108-38S4 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Vaccine; Human Papilloma Virus
Keywords: Adolescence; Attitudes; Parents; Vaccination
MeSH Terms: conditions — Behavior | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of which arm of social messaging they are receiving and whether they are receiving the control message or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Messaging (Experimental): Subjects are randomized to receive one of five messages on one of the four themes about HPV vaccination.
  Interventions: Other: Social Media Message about HPV and HPV vaccine
- Control Message (Other): Subjects are randomized to receive one of five messages about electronic cigarettes.
  Interventions: Other: Social media message about risk of electronic cigarettes.

INTERVENTIONS:
Other: Social Media Message about HPV and HPV vaccine — Messages educate parents with facts about HPV vaccination.
  Arms: HPV Messaging
Other: Social media message about risk of electronic cigarettes. — Messages educate parents with facts about electronic cigarettes. This is an attention control group without outcomes obtained.
  Arms: Control Message

SUMMARY:
This project involves a social media campaign to increase parent's knowledge and acceptance of the HPV (human papillomavirus) vaccine. The current vaccine protects against nine types of HPV, including seven that are known to cause cancer. The Centers for Disease Control and Prevention (CDC) estimates that the current HPV vaccine could prevent 90% of cancer cases caused by HPV, including cases of cervical cancer, oropharyngeal (mouth and throat) cancer, anal cancer, and others. About 150 and 104 cases of HPV-associated cancers are diagnosed each year in New Hampshire and Vermont, respectively-many of which could be prevented through vaccination. Currently, only 49.8% of New Hampshire adolescents and 44.3% of Vermont adolescents were not up-to-date for HPV vaccination as of 2016. This social media campaign is testing a set of campaign messages with parents locally and nationally to see which messages are most effective in improving their knowledge and acceptance of the vaccine. A study survey link will monitor the number of people reached and will measure parental intention to get their children vaccinated against HPV.

ELIGIBILITY:
Inclusion Criteria:

* parents of children 9-14 years old

Exclusion Criteria:

* non-parents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ardis L Olson, MD, Principal Investigator — Trustees of Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- See also: HPV cancer diagnosis rates — http://www.healthvermont.gov/sites/default/files/documents/pdf/stat_cancer_HPV_Assoc_Ca_Data_Brief.pdf
- See also: HPV vaccination rates — https://www.cdc.gov/mmwr/volumes/66/wr/mm6633a2.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1713 prospective participants responded to a social media or MTurk posting about the study between 12/12/18 to 04/15/19. 39 declined to consent. Of the remaining 1674 participants: 631 had no child and were deemed ineligible,.1043 people were eligible and consented to be in the study. Of that, 45 dropped before random assignment. As such, 998 people were eligible, provided a consent, and completed a baseline survey.
Pre-assignment Details: Eligible, consented participants completed a pre-test survey prior to assignment to an arm.
Groups:
- HPV Messaging: 834 Subjects were randomized to receive an experimental message about HPV vaccination.
- Control Messaging: 164 Subjects received a control message.
Period: Overall Study
Arm/Group | HPV Messaging | Control Messaging
Started | 834 | 164
Completed | 833 | 162
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: 1,713 participants initially recruited but 631 ineligible because no child leaving 1,043 eligible. Of eligibles 998 completed baseline survey.
Groups:
- HPV Messaging: 834 Subjects are randomized to receive one of five messages on one of the five themes about HPV vaccination.(165-167/group)
  Social Media Message about HPV and HPV vaccine: Messages educate parents with facts about HPV vaccination.
- Control Message: 164 Subjects are randomized to receive one of five messages about electronic cigarettes.
  Social media message about risk of electronic cigarettes.: Messages educate parents with facts about electronic cigarettes. This is an attention control group without outcomes obtained.
- Total: Total of all reporting groups
Arm/Group | HPV Messaging | Control Message | Total
Number analyzed (Participants) | 834 | 164 | 998
Age, Continuous [Mean (Standard Deviation); unit: years] — Years of age of parent as reported by study participant who identifies them as a parent on survey.
  years | 38.05 (10.75) | 37.33 (10.88) | 37.93 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 520 | 96 | 616
  Male | 314 | 68 | 382
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Prior knowledge of HPV [Count of Participants; unit: Participants] | 730 | 142 | 872
HPV Vaccine in prevents Cervical Cancer [Mean (Standard Deviation); unit: units on a scale] — This is a single question with the results reported as the answer from 1 to 5 on perceived effective of vaccine in preventing the cancer. Lower scores show a higher perception of it being effective. The full title is used without abbreviation.
  units on a scale | 2.53 (1.58) | 2.48 (1.50) | 2.52 (1.56)
HPV Vaccine in prevents Throat Cancer [Mean (Standard Deviation); unit: units on a scale] — 5 point scale from strongly disagree to strongly agree.
  This is a single question with the results reported as the answer from 1 to 5 on perceived effective of vaccine in preventing the cancer. Lower scores show a higher perception of it being effective. The full title is used without abbreviation.
  units on a scale | 2.26 (1.80) | 2.08 (1.81) | 2.23 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Change in Attitudes About HPV Vaccine
Description: Change in Attitudes about HPV vaccine: Pre to post test comparison of summated 9 items measured on a 7-point scale of HPV vaccine attitudes. Scores range from a minimum of 9 to a maximum of 63. Higher scores indicated more positive attitudes toward HPV vaccination. Change was calculated from two time points, the later time point(<1 hour post messaging intervention) minus value at baseline.
Time Frame: Post test completed < 1 hour post messaging intervention
Population: 1 participant in the experimental group and 2 participants in the control group withdrew from the study and are not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- HPV Messaging: 834 Subjects were randomized to receive one of 25 experimental messages about HPV vaccination
- Control Messaging: 164 Subjects received a control message not about HPV vaccination.
Arm/Group | HPV Messaging | Control Messaging
Number analyzed (Participants) | 833 | 162
units on a scale | .16 (.92) | -.08 (.91)
Statistical Analysis 1: Comparison: HPV Messaging vs Control Messaging; Test type: Superiority; p = .003, t-test, 2 sided

2. Secondary Outcome: Behavioral Intention to Vaccinate Their Child With HPV Vaccine
Description: A sub-group of parents of 9-14 year old children who had not been vaccinated were asked on pre- and post-test: How likely is it that she/he will receive the HPV vaccine in the next 12 months? Responses range form 1 (very likely) to 5 (not very likely).
  HPV vaccination behavioral intent change scores were calculated by subtracting pre- and post- test values. It is a negative-value scale, in which smaller values indicate more positive attitude change after exposure to the viewed message.
Time Frame: Ore test immediately before viewing message and post- test immediately after viewing message. Approximately one hour.
Population: A sub-group of parents of 9-14 year old children who had not been vaccinated were asked on pre- and post-test: How likely is it that she/he will receive the HPV vaccine in the next 12 months? Responses range form 1 (very likely) to 5 (not very likely).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- HPV Messaging: Subjects were randomized to receive one of 25 experimental messages about HPV vaccination.
  Behavioral intention to vaccinate only asked of the 155 HPV messaginglgroup parents with children 9-14 years who had not vaccinated their children at time of this experiment
- Control Message: Subjects received a control message not about HPV vaccination.
  Behavioral intention to vaccinate only asked of the 34 HPV controllgroup parents with children 9-14 years who had not vaccinated their children at time of this experiment
Arm/Group | HPV Messaging | Control Message
Number analyzed (Participants) | 155 | 34
units on a scale | -.022 (.81) | -.06 (.92)
Statistical Analysis 1: Comparison: HPV Messaging vs Control Message; Change in mean scores for behavioral intent to vaccine: negative values: smaller values indicate more likely to vaccinate; Test type: Superiority; p > .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events not anticipated over the < 1 hour of the study for a participant which only collects survey data about views of HPV vaccine
Description: Adverse events not collected
Arm/Group | HPV Messaging | Control Message
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03747302/Prot_SAP_000.pdf
  • Informed Consent Form: Phase 3 (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03747302/ICF_001.pdf
  • Informed Consent Form: Phase 2 (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT03747302/ICF_002.pdf